CLINICAL TRIAL: NCT01134770
Title: Prenatal Cocaine and Neurobehavioral Factors Underlying Mother-Infant Interaction
Brief Title: Prenatal Exposure Effects Psychophysiology Study
Acronym: PEEPS
Status: Enrolling by invitation | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: 08-1092
Record Dates: First submitted 2010-05-28; First posted 2010-06-02 (Estimated); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Pregnancy
Keywords: Prenatal Substance Use; Cocaine; Cigarette Smoking; Mothers; Pregnant women; Smoking Mothers
MeSH Terms: conditions — Cigarette Smoking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Plasma from mothers and buccal cells from infants will be stored for possible DNA analysis of target genes pending additional funding.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Prenatal Cocaine: Use of cocaine at anytime during pregnancy. Subjects may also have used other drugs in combination with Cocaine
- Prenatal Nicotine-Alcohol-Marijuana: Subjects may have used any of these drugs during pregnancy, alone or in combination. This group has not used cocaine during pregnancy.
- Drug-Free Pregnancy: Subjects did not use any of the following drugs during pregnancy:
  cocaine, nicotine, alcohol, marijuana.

SUMMARY:
The purpose of the study is to understand the biology and behavior of early mother-infant attachment, and to investigate how it may be affected by prenatal substance exposures. The investigators are interested in how drugs such as cocaine, alcohol, marijuana and cigarette smoking affect both mother and baby.

DETAILED DESCRIPTION:
The investigators are looking for pregnant women or mothers with their newborn infants to participate in this study. Eligible women include mothers who have used any of the following drugs at any time during pregnancy (alone or in combination):

1. cocaine
2. nicotine (cigarettes)
3. marijuana
4. alcohol

The investigators are also looking for mothers who have not used any drugs during pregnancy.

Information collected in this research study is strictly confidential, and protection of sensitive information is additionally assured by an NIH Certificate of Confidentiality.

Participation in this study involves:

1. One visit at 2-4 weeks postpartum. This visit includes an interview for mother and a 30 minute brain scan (no radiation, no sedation) for baby.
2. Two visits at 3 months postpartum. Mothers will have blood pressure and heart rate measured while they look at videos about babies, listen to baby sounds, interact with their own baby. Samples of blood, urine and saliva will be taken from mother. Baby will have a developmental assessment, and saliva samples will be taken.

Payment is $300 or the equivalent in Walmart gift cards for completion of brain imaging, lab visits and 1 day of monitoring mother's blood pressure at home.

ELIGIBILITY:
Inclusion Criteria:

* During pregnancy, mother has used any of the following:

  * cocaine
  * marijuana and/or alcohol but not cocaine
  * nicotine (smoked cigarettes)
  * no drugs during pregnancy
* Mother is pregnant or no more than 4 weeks postpartum

Exclusion Criteria:

* Mother has cardiovascular disease
* Delivery before 36 weeks or later than 42 weeks gestation
* Birth weight less than 5.5 lbs
* Baby was a multiple birth

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women or mothers with their newborn infants.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2008-07 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Determine the effect of prenatal cocaine exposure on the neonatal brain. ventricular volumes | 2 to 4 weeks of age

CONTACTS AND LOCATIONS:
Overall Officials: Karen Grewen, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No